CLINICAL TRIAL: NCT03884491
Title: Interventional, Open-label, Sequential-period Study Investigating the Pharmacokinetic Properties and Safety and Tolerability of Sublingual Formulations of Vortioxetine in Healthy Subjects
Brief Title: A Study Investigating Formulations of Vortioxetine Applied Under the Tongue in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18026A
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vortioxetine (Experimental)
  Interventions: Drug: Vortioxetine IV; Drug: Vortioxetine SLA; Drug: Vortioxetine SLB; Drug: Vortioxetine SLC

INTERVENTIONS:
Drug: Vortioxetine IV — an intravenous (IV) 10 mg dose (1 mg/mL) of vortioxetine infused over 2 hours
Drug: Vortioxetine SLA — 5-25 mg of sublingual formulation A of vortioxetine
Drug: Vortioxetine SLB — 5-25 mg of sublingual formulation B of vortioxetine
Drug: Vortioxetine SLC — formulation SLC: solution of vortioxetine, concentrate (12.5 mg/mL-62,5 mg/mL) 200 uL or 400 uL, SL, 5-25 mg

SUMMARY:
This study investigates formulations of vortioxetine applied under the tongue

DETAILED DESCRIPTION:
Apart from the first two doses, the study design is flexible in terms of doses and pharmaceutical formulations and will be decided upon based on an evaluation of the safety and tolerability as well as plasma exposure obtained during the study.

* The study consists of 5 periods. Single-doses of vortioxetine will be administered in all periods.
* All subjects will receive the same pharmaceutical formulations of the same dose strength in the same period and sequence.
* In Period 1, each subject will receive an intravenous (IV) 10 mg dose of vortioxetine infused over 2 hours. The exposure obtained after IV administration will serve as the reference for the sublingually administered dosage forms.
* In Period 2, each subject will receive 5 mg of formulation A (SLA) of vortioxetine in a sublingual (SL) formulation with a holding time of 90 seconds. The holding time is the time where swallowing of saliva should be avoided.
* For the 3 remaining dosing periods, one or more of the following options in pharmaceutical formulation, dose, and dosing condition apply to this study:

  * Increases or decreases in dose (≤25mg) using same formulation
  * Change from formulation SLA to formulation SLB
  * Change in the holding time
  * Change to formulation SLC
  * Change in swallowing technique of the sublingual dosage forms

ELIGIBILITY:
Inclusion Criteria:

-The subject has a BMI ≥18.5 and ≤30.0 kg/m2 at the Screening Visit and at the Baseline Visit.

Exclusion Criteria:

-The subject is identified or confirmed to be a CYP2D6 poor metabolizer (PM)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
absolute bioavailability (F) | From predose to 72 hours post dose
  absolute bioavailability of vortioxetine for the sublingual administrations
tmax | From predose to 72 hours post dose
  time to maximum plasma concentration (tmax)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- Quotient Sciences Ltd, Nottingham, United Kingdom